CLINICAL TRIAL: NCT06391008
Title: Immunosensitized Radiotherapy Combined With Evoximab (AK112) and Chemotherapy Neoadjuvant Therapy for Stage II-III Non-small Cell Lung Cancer: a Single Arm, Open Label, Phase II Clinical Study
Brief Title: Immunosensitized Radiotherapy Combined With Evoximab (AK112) and Chemotherapy Neoadjuvant Therapy for Stage II-III Non-small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SBRT-AK112-C
Record Dates: First submitted 2024-04-25; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Stereotactic Radiotherapy; Evoximab (AK112); New Adjuvant Therapy for Non-small Cell Lung Cancer
MeSH Terms: interventions — Radiosurgery; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT+Evoximab +pemetrexed/albumin paclitaxel+carboplatin (Experimental): Radiotherapy induction sensitization stage: For the primary lung lesion and irradiable mediastinal lymph nodes, stereotactic large segment radiotherapy is performed to complete the prescribed dose, PTV (planned target area): 5Gy x 3f.
  Drug combination therapy stage: Within 7 days after radiotherapy.Evoximab (20mg/kg, Q3W)+pemetrexed (500mg/m2, Q3W)/albumin paclitaxel 260 mg/m2, Q3W+carboplatin (AUC5, Q3W)
  Interventions: Radiation: Stereotactic radiotherapy; Drug: Evoximab; Drug: Pemetrexed; Drug: Albumin Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Radiation: Stereotactic radiotherapy — Targeting primary lung lesions and irradiable mediastinal lymph nodes, stereotactic large segment radiotherapy was performed to complete the prescribed dose, PTV (planned target area): 5Gy x 3f
Drug: Evoximab — Evoximab (20mg/kg, Q3W)
  Other Names: AK112
Drug: Pemetrexed — Pemetrexed (500mg/m2, Q3W)
Drug: Albumin Paclitaxel — Albumin Paclitaxel 260 mg/m2, Q3W
Drug: Carboplatin — Carboplatin (AUC5, Q3W)

SUMMARY:
This is an open label, prospective, single center Phase II clinical study. Intended to evaluate the main pathological response rate (MPR) and safety of stereotactic immunosensitized radiotherapy combined with Evoximab (PD-1/VEGF-A bispecific antibody) and chemotherapy neoadjuvant therapy for stage II-III NSCLC. Simultaneously observe and evaluate the complete pathological response rate (pCR), R0 resection rate, and event free survival (EFS) of stage II-III NSCLC treated with stereotactic radiotherapy combined with Evoximab (PD-1/VEGF-A bispecific antibody) and chemotherapy. Exploratory analysis based on serum/tumor molecular biological markers, as well as the optimal response time and mechanism for combined response.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined this study and signed an informed consent form;
2. ≥ 18 years old, both male and female are eligible;
3. Pathologically confirmed stage II-III NSCLC (AJCC 8th)
4. NSCLC confirmed by histology or cytology; No known EGFR/ALK gene mutations
5. ECOG score: 0-1;
6. Expected survival time ≥ 12 weeks;
7. The functions of important organs meet the following requirements:

   Absolute neutrophil count ≥ 1.5 × 10 ^ 9/L; Absolute lymphocyte count ≥ 0.8 × 10 ^ 9/L; Platelets ≥ 80 × 10 ^ 9/L; Hemoglobin ≥ 90g/L; Bilirubin ≤ 1.5 × ULN (within 7 days before the first medication); ALT and AST ≤ 1.5 × ULN (within 7 days before the first medication); Serum creatinine ≤ 1.5 × ULN;
8. Thyroid stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously, and if FT3 and FT4 levels are normal, they can be included in the study);
9. Non surgical sterilization or female patients of childbearing age are required to use a medically recognized contraceptive measure (such as an intrauterine device, contraceptive pill, or condom) during the study treatment period and within 3 months after the end of the study treatment period; Non surgically sterilized female patients of childbearing age must have a negative serum or urine HCG test within 72 hours prior to enrollment in the study; And it must be non lactation period; For male patients whose partners are women of childbearing age, effective methods of contraception should be used during the trial period and within 3 months after the last treatment medication.
10. Agree to provide blood samples and histological specimens. -

Exclusion Criteria:

1. The patient has any active autoimmune diseases or a history of autoimmune diseases (such as but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism; the patient has vitiligo; asthma that has completely relieved in childhood and does not require any intervention in adulthood can be included; asthma that requires medical intervention with bronchodilators cannot be included);
2. The patient is currently using immunosuppressive agents or systemic hormone therapy to achieve immunosuppressive effects (dosage>10mg/day prednisone or other therapeutic hormones), and continues to use them within 2 weeks prior to enrollment;
3. Has experienced severe allergic reactions to other monoclonal antibodies;
4. Suffering from hypertension and unable to achieve good control through antihypertensive drug treatment (systolic blood pressure ≥ 140mmHg or diastolic blood pressure ≥ 90mmHg);
5. There are clinical symptoms or diseases of the heart that cannot be well controlled, such as:

   NYHA grade 2 or above heart failure; Unstable angina pectoris; Have experienced myocardial infarction within one year; Clinically significant supraventricular or ventricular arrhythmias require treatment or intervention; QTc>450ms (male); QTc>470ms (female);
6. Abnormal coagulation function (INR>2.0, PT>16s), with a tendency to bleed or undergoing thrombolysis or anticoagulation treatment, allowing prophylactic use of low-dose aspirin and low molecular weight heparin;
7. Received previous anti-tumor immunotherapy, chemotherapy, and anti-tumor vaccine treatment (excluding adjuvant chemotherapy, if receiving adjuvant chemotherapy, disease recurrence or metastasis occurs more than 6 months after the last chemotherapy).
8. The patient has active infection, unexplained fever ≥ 38.5 ° C within 7 days before medication, or baseline white blood cell count>15 × 109/L; Individuals with purulent and chronic infections, and wounds that persist and do not heal;
9. Patients with bone metastases who have received palliative radiotherapy within the 4 weeks prior to participating in this study have a bone marrow area greater than 5%;
10. The patient has previously received anti PD-1, anti PD-L1, and anti PD-L2 treatments;
11. Individuals who are known to be allergic to the components of recombinant humanized anti-PD-1 monoclonal antibody drugs and vaccines;
12. Pregnant or lactating women, or female patients who have fertility but have not taken contraceptive measures;
13. Other malignant tumors (excluding basal cell or squamous cell carcinoma, superficial bladder cancer cancer, cervical carcinoma in situ or breast cancer) in the past 5 years;
14. Patients participating in other clinical trials simultaneously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Pathological Response (MPR) Rate | Up to 6 months
  MPR refers to pathology where the proportion of cancer cells in excised tumors and lymph nodes is less than 10%.
Safety and tolerability | Up to 6 months
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Pathological complete response (pCR) | Up to 6 months
  Pathological complete response (pCR): defined as the absence of residual tumor cells after evaluation of the excised tumor tissue and regional lymph nodes
EFS | Up to 6 months
  Event free survival (EFS): EFS is defined as the time from randomization to exclusion of surgical progression, local or distant recurrence, or death from any cause

OTHER OUTCOMES:
Exploratory purposes | Up to 6 months
  Exploratory analysis based on serum/tumor molecular biological markers, as well as the optimal response time and mechanism for combined response.

IPD SHARING:
Plan to Share IPD: No